CLINICAL TRIAL: NCT04077775
Title: Lumbopelvic Biomechanical Variables and TMJ Kinematics Changes in Pregnant Women: A Case-Control Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, rovan mohamed saad elbesh, Doctor, Misr University for Science and Technology
Other Study IDs: P.T.REC/012/001888
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Pelvic Pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study group (group A):: Study group (group ) Diagnostic Test: Study group (group A)24 women who have cyclic CPP
  I) Pelvic tilt angle:
  The physiotherapist stood beside the women and found the position of the anterior superior iliac spine (ASIS) and posterior superior iliac spine (PSIS) accurately while the woman was in standing position. Hence the therapist placed one end arm of PALM inclinometer on ASIS, and the other end arm was placed on PSIS. The pelvic sagittal inclination angle was the angle between the horizontal line and a line passing through the ASIS and PSIS that determined by the bubble level in the PALM inclinometer
  Interventions: Diagnostic Test: assesment
- Study group(group B):: included 20 women who have non-cyclic CPP and the other 16 women of the participants were normal I)
  Pelvic tilt angle:
  The physiotherapist stood beside the women and found the position of the anterior superior iliac spine (ASIS) and posterior superior iliac spine (PSIS) accurately. In contrast, the woman was in a standing position. Hence the therapist placed one end arm of PALM inclinometer on ASIS, and the other end arm was placed on PSIS. The pelvic sagittal inclination angle was the angle between the horizontal line and a line passing through the ASIS and PSIS that determined by the bubble level in the PALM inclinometer
  Diagnostic Test: Study group (group A)
- Control group (group C):: 16 women of the participants were normal and considered the control group
  I) Pelvic tilt angle:
  The physiotherapist stood beside the women and found the position of the anterior superior iliac spine (ASIS) and posterior superior iliac spine (PSIS) accurately while the woman was in standing position. Hence the therapist placed one end arm of PALM inclinometer on ASIS, and the other end arm was placed on PSIS. The pelvic sagittal inclination angle was the angle between the horizontal line and a line passing through the ASIS and PSIS that determined by the bubble level in the PALM inclinometer

INTERVENTIONS:
Diagnostic Test: assesment — assesment
  Groups: Study group (group A):

SUMMARY:
The relationship between the pelvis and stomatognathic system:

Various rationales for the relationship between the spine or pelvis and TMJ have been found. These theories include fascial, myological interrelationships, referred pain patterns and facilitating tonic neck reflexes involving inter segmental spinal pathways. A contributing mechanism could be the relationship between how TMJ occlusion, head position and body posture relate to the body's natural neurological visual/vestibular righting mechanism (Blum, 2004).

There is a Correlation between the facial axis together with the lordotic angle and the pelvic inclination, the inner gonial angle and the mandibular plane with the lordotic angle and the pelvic inclination, as well as the facial depth with the pelvic inclination showed a significant correlation (Carsten et al., 2007).

ELIGIBILITY:
Inclusion Criteria:

* The age of the participants will be ranged from 20 to 40 years. Their body mass index will be ranged from 20 to 25 kg/m2. They will have regular menstrual cycle. They will not receive any hormonal therapy or taking any regular drugs.

Exclusion Criteria:

* Bone disease. Discogenic state with radiculopathy or not. Systemic disease of musculoskeletal system. Any sensory problems. Previous vertebral fractures. Major spinal structural abnormality. Major jaw abnormality. Any jaw orthotics or prosthesis. Missing teeth.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: 30 women will participate in this study, thirty women diagnosed as having cyclic pelvic pain and thirty women diagnosed as having non cyclic pelvic pain thirty women normal women will not having pelvic pain. They will be selected from outpatient clinic of obstetrics and Gynaecology department in El-Hosary family health Centre.
  All participants will be given a full explanation of the protocol of the study and informed consent form will be signed from each subject before participating in the study
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
body mass index | 3 months
  BMI in kg/m^2
Satisfaction assessed by the VAS | 3 months
  Degrees of menstrual pain will be assessed using a VAS, which was a method of representing subjects' pain on a 10 cm linear scale. Score of 0 meant 'no pain' and 10 meant 'worst pain'. Tomeasure specific symptoms, such as the s
pelvic tilt in degrees: | 3 months
  The blocks are released and the rods are placed over the crest of the ilium. The blocks are then pressed firmly toward the midline. Read the angle from the level. If the gauge reads over 21/2°, the result is listed as positive.Anterior pelvic tilting angle: PALM was used for measuring pelvic tilting angle. A mark was put on a point just inferior to ASIS; another mark was put just inferior to PSIS. The callipers of the PALM were put on these two points
jaw movement | 3 months
  Maximal vertical mouth opening (MIO):
  From sitting position, with the use of the calliper, the distance between the incisal edges along the midline of the upper and lower central incisors without pain was measured, by placing one end of the poley gauge against the incisal edge of one of the upper central incisors, and the other end against the incisal edge of the opposing lower incisor.
  The distance recorded in millimeters, the subjects was instructed to" open your mouth as wide as possible without causing pain or discomfort". The poley gauge was sterilized with antiseptic solution before and after each measure
Spinal curves Measurement | 3 months
  spinal inclinations

CONTACTS AND LOCATIONS:
Locations (1):
- Rovan Elbesh, Giza, Egypt